CLINICAL TRIAL: NCT04618081
Title: Revlimid® Capsules General Drug Use-results Survey (Relapsed or Refractory Follicular Lymphoma and Marginal Zone Lymphoma)
Brief Title: Revlimid® Capsules General Drug Use-results Surveillance (Relapsed or Refractory FL and MZL)
Status: Completed | Type: Observational
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Other Study IDs: CC-5013-TCL-003; U1111-1260-3127 (Registry Identifier: WHO)
Record Dates: First submitted 2020-10-31; First posted 2020-11-05 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Lymphoma Nonhodgkin
Keywords: Lymphoma; Nonhodgkin; low-grade; B-cell; Follicular; Marginal zone; Safety; Revlimid; Rituximab; Actual use conditions; R2 combination therapy; Bone marrow depression; Neutropenia; Tumor flare
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma; Bone Marrow Failure Disorders; Neutropenia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with FL or MZL: Patients who have been diagnosed with follicular lymphoma (FL) or marginal zone lymphoma (MZL) who receive R2 combination therapy with revlimid and rituximab for the first time.

SUMMARY:
To ascertain the safety of Revlimid® Capsules 2.5 mg or 5 mg under the actual use conditions in patients who received R2 combination therapy with the drug and rituximab for the first time for relapsed or refractory follicular lymphoma (FL) or marginal zone lymphoma (MZL).

In particular, this surveillance will collect only information of occurrence state and treatment methods on bone marrow depression (neutropenia), which is specified as a safety specification, as well as on tumor flare, for which attention should be called.

1. Planned registration period 1.5 years
2. Planned surveillance period 3 years from the start of this survey

ELIGIBILITY:
Inclusion Criteria:

- Relapsed or Refractory Follicular Lymphoma or Marginal Zone Lymphoma

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This survey will be conducted in patients who have been diagnosed with follicular lymphoma (FL) or marginal zone lymphoma (MZL) who receive R2 combination therapy with the drug and rituximab for the first time.
Sampling Method: Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2020-12-17 (Actual); Primary Completion 2025-03-27 (Actual); Study Completion 2025-03-27 (Actual)

PRIMARY OUTCOMES:
Adverse Events (AEs) | Up to approximately 3 years
  Number of participants with adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Japan, Japan

IPD SHARING:
Plan to Share IPD: Yes
Information relating to our policy on data sharing and the process for requesting data can be found at the following link:
  https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/